CLINICAL TRIAL: NCT06723184
Title: Investigation of The Impact of Education Given to Grandmothers on Their Self-Confidence in Baby Care and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Busra nur Kutlu, Graduate student, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-60116787-020-468763
Record Dates: First submitted 2024-10-14; First posted 2024-12-09 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Voluntarily Accepting to Participate in the Study; At Least Primary School Graduate; Willing to Have Grandchildren or Having Grandchildren; Not Diagnosed With Any Psychiatric Illness
Keywords: Grandmother education; Grandchild care; Sense of self-confidence

STUDY DESIGN:
Intervention Model Description: Single blind pre-post test randomized controlled design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental grup (Experimental): Experimental grup
  Interventions: Behavioral: The training
- Control group (No Intervention): No intervention grup

INTERVENTIONS:
Behavioral: The training — Behavioral: Antenatal Education Education Hours: The training will be completed in a total of three weeks and six hours, two hours each week.
  Method: The training will be in a total of three weeks and six hours, two hours each week. "Informed Voluntary Consent Form" will be obtained from individuals in both groups. Grandmothers in both the control and intervention groups will be asked to fill out the "Introductory Information Form, Pharis Self-Confidence Scale, State-Trait Anxiety Scale and Knowledge Measurement Questionnaire for Grandchild Care" measurement tools. The data of the intervention group will be filled in before and after the training. The data of the control group will be filled in parallel with the intervention group. At the end of the study, the same training will be applied to the control group.
  Group to receive training: Grandmothers who are expecting a grandchild and have a grandchild will be included in the training.
  Arms: Experimental grup

SUMMARY:
Although there are studies in the literature on the effects of antenatal education on pregnant women, there are no interventional studies on the education of grandmothers, who play an important role in the care of the newborn baby. Therefore, the aim of this study is to examine the effects of antenatal education given to grandmothers on anxiety and self-confidence in baby care. The type of study is a randomized controlled experimental study with pre-post and control groups. The training will be given face to face to grandmothers reached through social media. At the beginning of the study, the sample size was calculated in the G-Power program by taking as reference a similar study in which the same scale (Pharis Self-Confidence Scale) was used. According to the t-test in independent groups, 95% confidence interval, 95% power and high effect size (0.98), a total of 48 people were required, 24 experimental and 24 control. Women who apply to receive training will be assigned to intervention and control groups in a block randomised manner according to their application numbers. Intention-to-treat analysis will be performed to prevent bias and losses. A total of six hours of training will be provided to the intervention group. The program content will be prepared by researchers based on literature and using childbirth preparation education philosophies.

DETAILED DESCRIPTION:
The research is a randomized controlled experimental study with a pre-test-post-test control group. The research will be conducted with women who are grandmothers. At the beginning of the study, the sample size was calculated in the G-Power program by taking as reference a similar study in which the same scale (Pharis Self-Confidence Scale) was used. According to the t-test in independent groups, 95% confidence interval, 95% power and high effect size (0.98), a total of 48 people were required, 24 experimental and 24 control. Participants will be reached via social media. In this study, the Introductory Information Form, Pharis Self-Confidence Scale, State-Trait Anxiety Scale and Grandchild Care Knowledge Measurement Questionnaire, which reflect the sociodemographic characteristics of the participants, will be used. Women who apply with the request to receive training will be assigned to the intervention and control groups in a block randomization according to their application numbers. Intention-to-treat analysis will be performed to prevent bias and losses. As the randomization method, "block randomization" will be used to ensure that the sample size is equal in the study and control groups. Randomization will be done using the www.randomizer.org application. Data will be analyzed using the SPSS (23.0) package program. Alpha 0.05 will be accepted for significance. Mann Whitney U test and Chi-Square tests will be used to determine whether there is a difference between the groups in terms of demographic variables. Mann Whitney U test will be used to determine the difference between the Pharis Self-Esteem Scale and State-Trait Anxiety Inventory scale scores between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily accepting to participate in the study
* At least primary school graduate
* Willing to have grandchildren or having grandchildren
* Not diagnosed with any psychiatric illness

Exclusion Criteria:

* Not willing to participate in the study
* Not having at least a primary school degree
* Being diagnosed with a psychiatric disorder
* Not having grandchildren or not having grandchildren

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Willing to have grandchildren or having grandchildren
Enrollment: 48 (Actual)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | It will be applied to both the experimental and control groups within 3 days before the training.
  This form, created in line with the literature, consists of 9 questions that include some socio-demographic characteristics of grandmothers.
Knowledge Measurement Survey for Grandchild Care | It will be applied to both the experimental and control groups within 3 days before the training.
  This survey will be used to measure the knowledge level of grandmothers on topics parallel to the training content to be created and the effectiveness of the planned training. The survey consists of 25 questions.
State and Trait Anxiety Scale | It will be applied to both the experimental and control groups within 3 days before the training.
  The scale was developed by Spielberger et al to determine state and trait anxiety levels separately . The Turkish adaptation of the form was made by Öner et al. The Cronbach Alpha value of the State Anxiety Scale was found to be between 0.83-0.87, and the Cronbach Alpha value of the Trait Anxiety Scale was found to be between 0.94-0.96. The inventory has two separate scales, each consisting of 20 items:
  1. State Anxiety Scale: Determines how the individual feels at a certain moment and under certain conditions.
  2. Trait Anxiety Scale: Determines how the individual generally feels, regardless of the situation and conditions they are in.
Pharis Self-Confidence Scale | It will be applied to both the experimental and control groups within 3 days before the training.
  First developed by Pharis and later by Walker the internal consistency reliability was found to be between 71-91 in a study. In 2003, the validity reliability in Turkey was made by Hüsniye Çalışır. The Pharis self-confidence scale, a 13-item five-point measurement tool, measures a parent's own feelings of confidence about daily baby care. Each baby care item is rated from one (not at all) to five (completely). A high score indicates high self-confidence in baby care. The Cronbach alpha internal consistency coefficient of the scale was found to be 0.86

SECONDARY OUTCOMES:
Knowledge Measurement Survey for Grandchild Care | The scale will be applied to the experimental group within 3 days after the training, and to the control group at parallel times with the experimental group.
  This survey will be used to measure the knowledge level of grandmothers on topics parallel to the training content to be created and the effectiveness of the planned training. The survey consists of 25 questions.
State and Trait Anxiety Scale | The scale will be applied to the experimental group within 3 days after the training, and to the control group at parallel times with the experimental group.
  The scale was developed by Spielberger et al to determine state and trait anxiety levels separately . The Turkish adaptation of the form was made by Öner et al. The Cronbach Alpha value of the State Anxiety Scale was found to be between 0.83-0.87, and the Cronbach Alpha value of the Trait Anxiety Scale was found to be between 0.94-0.96. The inventory has two separate scales, each consisting of 20 items:
  1. State Anxiety Scale: Determines how the individual feels at a certain moment and under certain conditions.
  2. Trait Anxiety Scale: Determines how the individual generally feels, regardless of the situation and conditions they are in.
Pharis Self-Confidence Scale | The scale will be applied to the experimental group within 3 days after the training, and to the control group at parallel times with the experimental group.
  First developed by Pharis and later by Walker the internal consistency reliability was found to be between 71-91 in a study. In 2003, the validity reliability in Turkey was made by Hüsniye Çalışır. The Pharis self-confidence scale, a 13-item five-point measurement tool, measures a parent's own feelings of confidence about daily baby care. Each baby care item is rated from one (not at all) to five (completely). A high score indicates high self-confidence in baby care.The Cronbach alpha internal consistency coefficient of the scale was found to be 0.86

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University Faculty of Health Sciences, Denizli, Kınıklı, Turkey (Türkiye)